CLINICAL TRIAL: NCT00528086
Title: A Single Center, Randomized Controlled, Pilot Study Comparing Group Visits Versus Routine Clinical Care for Participants With Parkinson's Disease (PD).
Brief Title: A Pilot, Randomized Controlled Trial of Group Visits for Persons With Parkinson's Disease
Acronym: GROUP-PD
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Parkinson Foundation (Other)
Responsible Party: E. Ray Dorsey, MD, MBA, University of Rochester
Other Study IDs: RSRB00019885
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Parkinson's Disease; Parkinson's Disease Patient Caregivers
Keywords: Group visits
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Parkinson disease patients and their family members or caregivers randomly assigned to receive their PD care in group visit format.
- 2: Parkinson disease patients and their family members or caregivers randomly assigned to receive their PD care in standard of care format (one-on-one physician-patient visits).

SUMMARY:
To determine patient satisfaction with group visits versus standard of care delivery for patients with Parkinson's disease.

DETAILED DESCRIPTION:
To establish the feasibility and to estimate the benefit of group visits for individuals with PD and their caregivers. The feasibility will be assessed by the ability to enroll and retain (measured by number of individuals who complete the 12-month study and at least half the study visits) ~40 individuals in the pilot trial. The responsiveness of the following different outcomes to group visits will be assessed during the pilot trial: quality of life, patient satisfaction, depression, caregiver burden, resource utilization, and disease progression. The primary outcome measure for efficacy will be a comparison of the change in the Parkinson's Disease Questionnaire-39 from baseline to 12 months in the control (routine care) and intervention (group visit) groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease as determined by having two of the four cardinal features of PD (rest tremor, bradykinesia, cogwheel rigidity, and gait instability) and no alternative explanation for the etiology of the symptoms
* Willing and able to provide informed consent and to participate actively in group visits and complete study activities

Exclusion Criteria:

* Cognitive impairment, psychiatric disorder, or history of or current clinically significant substance abuse that in the investigator's judgment could interfere in the conduct of group visits or with study participation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from Drs. Dorsey, Biglan, and Marshall's patient populations from the Parkinson disease clinic at the University of Rochester Neurology group.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The feasibility (based on the ability to enroll and retain 40 individuals) and benefit (based on the 12-month change in PDQ-39) of group visits for individuals with Parkinson disease and their caregivers. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: E. Ray Dorsey, MD, MBA, Principal Investigator — University of Rochester; Kevin Biglan, MD, MPH, Principal Investigator — University of Rochester; Fred Marshall, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Beck A, Scott J, Williams P, Robertson B, Jackson D, Gade G, Cowan P. A randomized trial of group outpatient visits for chronically ill older HMO members: the Cooperative Health Care Clinic. J Am Geriatr Soc. 1997 May;45(5):543-9. doi: 10.1111/j.1532-5415.1997.tb03085.x. PMID 9158573
- [Background] Scott JC, Conner DA, Venohr I, Gade G, McKenzie M, Kramer AM, Bryant L, Beck A. Effectiveness of a group outpatient visit model for chronically ill older health maintenance organization members: a 2-year randomized trial of the cooperative health care clinic. J Am Geriatr Soc. 2004 Sep;52(9):1463-70. doi: 10.1111/j.1532-5415.2004.52408.x. PMID 15341547
- [Background] Masley S, Phillips S, Copeland JR. Group office visits change dietary habits of patients with coronary artery disease-the dietary intervention and evaluation trial (D.I.E.T.). J Fam Pract. 2001 Mar;50(3):235-9. PMID 11252212
- [Background] Coleman EA, Grothaus LC, Sandhu N, Wagner EH. Chronic care clinics: a randomized controlled trial of a new model of primary care for frail older adults. J Am Geriatr Soc. 1999 Jul;47(7):775-83. doi: 10.1111/j.1532-5415.1999.tb03832.x. PMID 10404919
- [Background] Trento M, Passera P, Tomalino M, Bajardi M, Pomero F, Allione A, Vaccari P, Molinatti GM, Porta M. Group visits improve metabolic control in type 2 diabetes: a 2-year follow-up. Diabetes Care. 2001 Jun;24(6):995-1000. doi: 10.2337/diacare.24.6.995. PMID 11375359
- [Background] Wagner EH, Grothaus LC, Sandhu N, Galvin MS, McGregor M, Artz K, Coleman EA. Chronic care clinics for diabetes in primary care: a system-wide randomized trial. Diabetes Care. 2001 Apr;24(4):695-700. doi: 10.2337/diacare.24.4.695. PMID 11315833
- [Background] Ickovics JR, Kershaw TS, Westdahl C, Rising SS, Klima C, Reynolds H, Magriples U. Group prenatal care and preterm birth weight: results from a matched cohort study at public clinics. Obstet Gynecol. 2003 Nov;102(5 Pt 1):1051-7. doi: 10.1016/s0029-7844(03)00765-8. PMID 14672486
- [Background] Grosset KA, Grosset DG. Patient-perceived involvement and satisfaction in Parkinson's disease: effect on therapy decisions and quality of life. Mov Disord. 2005 May;20(5):616-9. doi: 10.1002/mds.20393. PMID 15719417
- [Background] Shimbo T, Goto M, Morimoto T, Hira K, Takemura M, Matsui K, Yoshida A, Fukui T. Association between patient education and health-related quality of life in patients with Parkinson's disease. Qual Life Res. 2004 Feb;13(1):81-9. doi: 10.1023/B:QURE.0000015306.59840.95. PMID 15058790
- [Background] Global Parkinson's Disease Survey (GPDS) Steering Committee.. Factors impacting on quality of life in Parkinson's disease: results from an international survey. Mov Disord. 2002 Jan;17(1):60-7. doi: 10.1002/mds.10010. PMID 11835440
- [Background] Christakis NA, Allison PD. Mortality after the hospitalization of a spouse. N Engl J Med. 2006 Feb 16;354(7):719-30. doi: 10.1056/NEJMsa050196. PMID 16481639
- [Background] Aarsland D, Larsen JP, Karlsen K, Lim NG, Tandberg E. Mental symptoms in Parkinson's disease are important contributors to caregiver distress. Int J Geriatr Psychiatry. 1999 Oct;14(10):866-74. PMID 10521886
- [Background] Schrag A, Hovris A, Morley D, Quinn N, Jahanshahi M. Caregiver-burden in parkinson's disease is closely associated with psychiatric symptoms, falls, and disability. Parkinsonism Relat Disord. 2006 Jan;12(1):35-41. doi: 10.1016/j.parkreldis.2005.06.011. Epub 2005 Nov 3. PMID 16271496
- [Background] Schrag A, Jahanshahi M, Quinn N. What contributes to quality of life in patients with Parkinson's disease? J Neurol Neurosurg Psychiatry. 2000 Sep;69(3):308-12. doi: 10.1136/jnnp.69.3.308. PMID 10945804
- [Background] Slawek J, Derejko M, Lass P. Factors affecting the quality of life of patients with idiopathic Parkinson's disease--a cross-sectional study in an outpatient clinic attendees. Parkinsonism Relat Disord. 2005 Nov;11(7):465-8. doi: 10.1016/j.parkreldis.2005.04.006. Epub 2005 Sep 9. PMID 16154794
- [Background] Whetten-Goldstein K, Sloan F, Kulas E, Cutson T, Schenkman M. The burden of Parkinson's disease on society, family, and the individual. J Am Geriatr Soc. 1997 Jul;45(7):844-9. doi: 10.1111/j.1532-5415.1997.tb01512.x. PMID 9215336
- [Background] Noyes K, Liu H, Li Y, Holloway R, Dick AW. Economic burden associated with Parkinson's disease on elderly Medicare beneficiaries. Mov Disord. 2006 Mar;21(3):362-72. doi: 10.1002/mds.20727. PMID 16211621
- [Background] Peto V, Jenkinson C, Fitzpatrick R, Greenhall R. The development and validation of a short measure of functioning and well being for individuals with Parkinson's disease. Qual Life Res. 1995 Jun;4(3):241-8. doi: 10.1007/BF02260863. PMID 7613534
- [Background] Marinus J, Ramaker C, van Hilten JJ, Stiggelbout AM. Health related quality of life in Parkinson's disease: a systematic review of disease specific instruments. J Neurol Neurosurg Psychiatry. 2002 Feb;72(2):241-8. doi: 10.1136/jnnp.72.2.241. PMID 11796776
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Essink-Bot ML, Stouthard ME, Bonsel GJ. Generalizability of valuations on health states collected with the EuroQolc-questionnaire. Health Econ. 1993 Oct;2(3):237-46. doi: 10.1002/hec.4730020307. PMID 8275169
- [Background] Schrag A, Selai C, Jahanshahi M, Quinn NP. The EQ-5D--a generic quality of life measure-is a useful instrument to measure quality of life in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jul;69(1):67-73. doi: 10.1136/jnnp.69.1.67. PMID 10864606
- [Background] Escobar GJ, Braveman PA, Ackerson L, Odouli R, Coleman-Phox K, Capra AM, Wong C, Lieu TA. A randomized comparison of home visits and hospital-based group follow-up visits after early postpartum discharge. Pediatrics. 2001 Sep;108(3):719-27. doi: 10.1542/peds.108.3.719. PMID 11533342
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Ertan FS, Ertan T, Kiziltan G, Uygucgil H. Reliability and validity of the Geriatric Depression Scale in depression in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2005 Oct;76(10):1445-7. doi: 10.1136/jnnp.2004.057984. PMID 16170093
- [Background] Weintraub D, Moberg PJ, Duda JE, Katz IR, Stern MB. Effect of psychiatric and other nonmotor symptoms on disability in Parkinson's disease. J Am Geriatr Soc. 2004 May;52(5):784-8. doi: 10.1111/j.1532-5415.2004.52219.x. PMID 15086662
- [Background] Zarit SH, Todd PA, Zarit JM. Subjective burden of husbands and wives as caregivers: a longitudinal study. Gerontologist. 1986 Jun;26(3):260-6. doi: 10.1093/geront/26.3.260. No abstract available. PMID 3721233
- [Background] Elmstahl S, Ingvad B, Annerstedt L. Family caregiving in dementia: prediction of caregiver burden 12 months after relocation to group-living care. Int Psychogeriatr. 1998 Jun;10(2):127-46. doi: 10.1017/s1041610298005249. PMID 9677500
- [Background] Goetz CG, Stebbins GT. Risk factors for nursing home placement in advanced Parkinson's disease. Neurology. 1993 Nov;43(11):2227-9. doi: 10.1212/wnl.43.11.2227. PMID 8232934
- [Background] Fahn S, Oakes D, Shoulson I, Kieburtz K, Rudolph A, Lang A, Olanow CW, Tanner C, Marek K; Parkinson Study Group. Levodopa and the progression of Parkinson's disease. N Engl J Med. 2004 Dec 9;351(24):2498-508. doi: 10.1056/NEJMoa033447. PMID 15590952
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Montgomery GK, Reynolds NC Jr, Warren RM. Qualitative assessment of Parkinson's disease: study of reliability and data reduction with an abbreviated Columbia Scale. Clin Neuropharmacol. 1985;8(1):83-92. PMID 3978653
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Deuschl G, Schade-Brittinger C, Krack P, Volkmann J, Schafer H, Botzel K, Daniels C, Deutschlander A, Dillmann U, Eisner W, Gruber D, Hamel W, Herzog J, Hilker R, Klebe S, Kloss M, Koy J, Krause M, Kupsch A, Lorenz D, Lorenzl S, Mehdorn HM, Moringlane JR, Oertel W, Pinsker MO, Reichmann H, Reuss A, Schneider GH, Schnitzler A, Steude U, Sturm V, Timmermann L, Tronnier V, Trottenberg T, Wojtecki L, Wolf E, Poewe W, Voges J; German Parkinson Study Group, Neurostimulation Section. A randomized trial of deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Aug 31;355(9):896-908. doi: 10.1056/NEJMoa060281. PMID 16943402